CLINICAL TRIAL: NCT06903325
Title: A Prospective Multicentre Clinical Study of Dynamic Monitoring of Plasma ctDNA Methylation Markers to Predict Recurrence of Colorectal Cancer After Complete Resection of Peritoneal Metastases
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Guoxiang Cai, Professor, Fudan University
Other Study IDs: CRIP-ctDNA
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Peritoneal Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POM1 positive: Patients whose 1-month-postoperative plasma ctDNA methylation status is positive
  Interventions: Other: As an observational study, we did not intervene
- POM1 negative: Patients whose 1-month-postoperative plasma ctDNA methylation status is negative
  Interventions: Other: As an observational study, we did not intervene

INTERVENTIONS:
Other: As an observational study, we did not intervene — Interventions

SUMMARY:
The goal of this clinical trial is to explore the predictive effect of postoperative plasma ctDNA methylation status on postoperative recurrence free survival (RFS) of colorectal cancer patients with peritoneal metastasis after R0/R1 resection. The main questions it aims to answer are:

Preoperative and postoperative plasma ctDNA methylation detection (ColonAiQ) was performed in patients with peritoneal metastasis from colorectal cancer who underwent R0/R1 resection. Clinical information of patients was collected to explore the predictive effect of postoperative plasma ctDNA methylation status on postoperative recurrence free survival (RFS) of colorectal cancer patients with peritoneal metastasis.

Participants will:

The patients were followed up according to the normal review procedure of the hospital and the NCCN guidelines until at least 24 months after surgery. The review content included CT/MRI imaging evaluation and blood CEA (every 3 months). Whole-blood samples were obtained for timely plasma separation and ctDNA extraction at 1 month after surgery (before the start of postoperative chemotherapy) and every 3 months through 24 months after surgery. One blood sample was obtained when tumor recurrence was first detected on imaging.

Detection of methylation in tissue and plasma samples

1. GutSeer methylation NGS was performed on peritoneal metastatic cancer tissues and paired normal peritoneal tissues.
2. ctDNA GutSeer methylation NGS was performed on plasma samples before surgery, 1 month after surgery, 24 months after surgery, and when tumor recurrence was first detected by imaging examination.
3. ctDNA methylation PCR (ColonAiQ) was performed on plasma samples before surgery, 1 month after surgery, every 3 months to 24 months after surgery, and when tumor recurrence was first detected by imaging examination.

ELIGIBILITY:
Inclusion Criteria:

-1. No gender limit, age greater than 18 years old; 2, ECOG score ≤1; 3. Life expectancy ≥2 years; 4. Colorectal adenocarcinoma/mucinous adenocarcinoma/signet ring cell carcinoma confirmed by histopathology; 5, preoperative PCI score ≤20, peritoneal tumor cytoreductive surgery (CRS), surgery to achieve R0/1 resection; 6. Be able to understand the situation of this study and sign the informed consent.

7. The primary colorectal cancer has undergone R0 resection, and there is no extraperitoneal metastasis (except ovary).

Exclusion Criteria:

* 1. Combined with primary malignant tumors of other organs (current or within the past 5 years) (excluding patients with skin basal cell carcinoma and cervical carcinoma in situ undergoing radical treatment); 2. Severe mental illness or drug abuse; 3, severe heart, lung, vascular disease can not tolerate surgery; 4. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peritoneal metastasis from colorectal cancer whose preoperative imaging PCI score was ≤20 and could be evaluated for R0/R1 resection were screened for enrollment. Preoperative plasma samples and tumor tissue samples were collected for ctDNA multigene methylation markers detection. Patients who achieved R0/R1 resection of peritoneal carcinomatosis were enrolled in this clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
predictive value of ColonAiQ postoperative recurrence free survival (RFS) | 2023.10-2027.10
  explore the predictive effect of postoperative plasma ctDNA methylation status on postoperative recurrence free survival (RFS) of colorectal cancer patients with peritoneal metastasis.

SECONDARY OUTCOMES:
predictive value of GutSeer for RFS | 2023.10-2027.10
  Preoperative and postoperative plasma ctDNA polygene methylation test (GutSeer) was performed in patients with peritoneal metastasis from colorectal cancer who underwent R0/R1 resection, and the clinical information of patients' recurrence-free survival (RFS) was collected to explore the predictive effect of postoperative plasma ctDNA methylation status on postoperative RFS of colorectal cancer peritoneal metastasis.
predictive value of ctDNA for dynamic monitoring | 2023.10-2027.10
  To explore the predictive value of plasma ctDNA methylation status before surgery, after postoperative adjuvant chemotherapy, and regularly monitored after surgery for recurrence and metastasis of colorectal cancer patients with peritoneal metastasis
difference of predictive value of ColonAiQ and GutSeer | 2023.10-2027.10
  Compare the prognostic value of GutSeer and ColonAiQ and CEA at 1 month after surgery;
the advance time of dynamic detection of plasma ctDNA methylation compared with imaging monitoring | 2023.10-2027.10
  To explore the advance time of dynamic detection of plasma ctDNA methylation compared with imaging monitoring in monitoring recurrence after complete resection of peritoneal metastasis from colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Guoxiang Cai, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The results of clinical trials will be published in the form of a paper, but content involving patient personal information or sensitive information will be kept confidential as required by the Ethics Committee